CLINICAL TRIAL: NCT04340271
Title: The Clinical Utility of Extracorporeal Shock Wave Therapy on Burns of Upper Extremity : Controlled, Randomization, Double Bilind Study
Brief Title: The Clinical Utility of Extracorporeal Shock Wave Therapy on Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangang Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, So Young Joo, Clinical professor, Hangang Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HangangSHH-10
Record Dates: First submitted 2020-04-02; First posted 2020-04-09 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Burn Scar
Keywords: burn scar; extracorporeal shock wave therapy; skin characteristics
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: The patients' burn scars had re-epithelialized after split-thickness skin graft (STSG). We included patients aged ≥18 years with a deep partial-thickness (second-degree) burn or a full thickness (third-degree) burn to their upper extremities, having been transferred to the rehabilitation department after acute burn treatment, and less than 6 months since the onset of the burn injury.
Who Masked: Participant, Outcomes Assessor
Masking Description: 1. The patients didnot know whether it is included in the experimental group and control group
  2. Outcome measurements and data analyses were performed by a trained and blinded outcome assessor who was not involved in the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal shock wave therapy group (Experimental): Patients in the ESWT group were explained to select the most hypertrophic and retracting area for the treatment on dominant hand. ESWT was conducted using the Duolith SD-1® device (StorzMedical, Tägerwilen, Switzerland) with an electromagnetic cylindrical coil source for the focused shock wave (Fig. 2). ESWT was performed around the primary treatment site at 100 impulses/cm2, an energy flux density(EFD) of 0.05 to 0.30 mJ/mm2, frequency of 4Hz, and 1000 to 2000 impulses were administered at 1-week intervals for 4 sessions.
  Interventions: Other: Extracorporeal shock wave therapy; Other: conventional occupational therapy
- sham stimulation group (Sham Comparator): The same shock wave equipment used in the experimental group was used with a sham adapter that had the same shape but emitted no energy
  Interventions: Other: conventional occupational therapy

INTERVENTIONS:
Other: Extracorporeal shock wave therapy — ESWT was conducted using the Duolith SD-1® device (StorzMedical, Tägerwilen, Switzerland) with an electromagnetic cylindrical coil source for the focused shock wave (Fig. 2). ESWT was performed around the primary treatment site at 100 impulses/cm2, an energy flux density(EFD) of 0.05 to 0.30 mJ/mm2, frequency of 4Hz, and 1000 to 2000 impulses were administered at 1-week intervals for 4 sessions.
  Arms: Extracorporeal shock wave therapy group
Other: conventional occupational therapy — Standard accupational therapy consist of range of motion exercise, strengthening exercises, and activities of daily living exercises

SUMMARY:
In burn patients, the wound healing process may lead to a fibrotic hypertrophic scar, which is raised, inflexible and responsible functional impairments. There are few studies which have investigated the effect of extracorporeal shock wave therapy (ESWT) on hypertrophic scar characteristics using objective measurements. Thus, this study aimed to ascertain the effects of ESWT on burn scars using objective measurements. This double-blinded, randomized, controlled trial involved 36 patients with burns. Patients were randomized into a ESWT (an energy flux density (EFD) of 0.05 to 0.30 mJ/mm2, frequency of 4Hz, and 1000 to 2000 impulses) or a sham stimulation group.

DETAILED DESCRIPTION:
In burn patients, the wound healing process may lead to a fibrotic hypertrophic scar, which is raised, inflexible and responsible functional impairments. There are few studies which have investigated the effect of extracorporeal shock wave therapy (ESWT) on hypertrophic scar characteristics using objective measurements. Thus, this study aimed to ascertain the effects of ESWT on burn scars using objective measurements. This double-blinded, randomized, controlled trial involved 36 patients with burns. Patients were randomized into a ESWT (an energy flux density (EFD) of 0.05 to 0.30 mJ/mm2, frequency of 4Hz, and 1000 to 2000 impulses) or a sham stimulation group. Each intervention was applied to the hypertrophic scars of upper extremities after autologous split-thickness skin grafting (STSG) using Materiderm for 4 weeks once per week. The ESWT group (n=18) received shock waves with low-energy flux density (0.05-0.30 mJ/mm2). The interval between treatments is a 1-week. The ESWT group also received standard treatment. The control group (n=18) received sham stimulation with standard treatment. The investigators compared the skin quality of the ESWT and control groups. Participants were made comfortable and acclimatized to room conditions. Room temperature was maintained at 20-25'C and relative humidity at 40-50 %. In the supine position, skin properties were measured. The thickness was measured with a ultrasonic wave equipment (128 BW1 Medison, Korea). Mexameter® (MX18, Courage-Khazaka Electronics GmbH, Germany) was used to measure melanin levels and the severity of erythema. The higher values indicating a darker and redder skin. TEWL was measured with a Tewameter® (Courage-Khazaka Electronic GmbH, Germany), which is used for evaluating water evaporation. Sebum in the scars was measured with the Sebumeter® (Courage-Khazaka Electronic GmbH, Germany). The measurement is based on the principle of grease-spot photometry using a cassette with its special tape. A microprocessor calculates the result, which is shown on the display in mg/cm2. Elasticity was measured using Cutometer SEM 580® (Courage-Khazaka Electronic GmbH, Cologne, Germany), which applies negative pressure (450 mbar) on the skin. The numeric values (mm) of the skin's distortion is presented as the elasticity. Two seconds of negative pressure of 450 mbar is followed by 2 s of recess, and this consists of a complete cycle. Three measurement cycles were conducted, and the average values were obtained.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years
* deep partial-thickness (second-degree) burn or a full thickness (third-degree) burn
* less than 6 months since the onset of the burn injury

Exclusion Criteria:

* history of cancer
* fourth-degree burns (involving muscles, tendons, and bone injuries)
* musculoskeletal diseases (fracture, amputation, rheumatoid arthritis, and degenerative joint diseases)
* pregnancy
* if there was potential for additional damage to the skin due to the use of ESWT and conventional occupational therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
scar thickness | 4 weeks
  The thickness was measured with a ultrasonic wave equipment

SECONDARY OUTCOMES:
skin darkness | 4 weeks
  the degree of pigmentation and melanin level, the higher values indicating a darker(AU)
skin reddness | 4 weeks
  the degree of erythema, the higher values indicating a redder skin(AU)
skin dryness | 4 weeks
  evaluating the degree of water evaporation(g/h/m2). the higher values indicating a skin dryness
sebum level | 4 weeks
  measurement is based on the principle of grease-spot photometry using a cassette with its special tape. A microprocessor calculates the result, which is shown on the display in mg/cm2
Elasticity | 4 weeks
  which applies negative pressure (450 mbar) on the skin. The numeric values (mm) of the skin's distortion is presented as the elasticity. Two seconds of negative pressure of 450 mbar is followed by 2 s of recess, and this consists of a complete cycle. Three measurement cycles were conducted, and the average values were obtained

CONTACTS AND LOCATIONS:
Locations (1):
- Hangang Sacred Heart Hospital, Seoul, Yeong-deungpo-Dong, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cui HS, Hong AR, Kim JB, Yu JH, Cho YS, Joo SY, Seo CH. Extracorporeal Shock Wave Therapy Alters the Expression of Fibrosis-Related Molecules in Fibroblast Derived from Human Hypertrophic Scar. Int J Mol Sci. 2018 Jan 2;19(1):124. doi: 10.3390/ijms19010124. PMID 29301325
- [Result] Saggini R, Saggini A, Spagnoli AM, Dodaj I, Cigna E, Maruccia M, Soda G, Bellomo RG, Scuderi N. Extracorporeal Shock Wave Therapy: An Emerging Treatment Modality for Retracting Scars of the Hands. Ultrasound Med Biol. 2016 Jan;42(1):185-95. doi: 10.1016/j.ultrasmedbio.2015.07.028. Epub 2015 Oct 9. PMID 26454624